CLINICAL TRIAL: NCT01012440
Title: Role of PEM Flex Solo II PET Scanner in Evaluating Neoadjuvant Chemotherapy Response in Patients With Breast Cancer
Brief Title: Role of Positron Emission Mammography (PEM) Flex Solo II Positron Emission Tomography (PET) Scanner in Evaluating Neoadjuvant Chemotherapy Response in Patients With Breast Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor accrual
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16895A
Record Dates: First submitted 2009-06-25; First posted 2009-11-13 (Estimated); Results first posted 2015-07-27 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Beast cancer subjects (Experimental): Subject will have assessment of neoadjuvant chemotherapy treatment response by both MRI and PEM to compare methods
  Interventions: Device: PEM Flex Solo II PET Scanner; Device: MRI scan

INTERVENTIONS:
Device: PEM Flex Solo II PET Scanner — Subjects will receive bilateral (both sides) breast and axillary PEM scans.
Device: MRI scan — Subjects will receive bilateral (both sides) breast and axillary MRI scans.

SUMMARY:
The purpose of this study is:

1. To evaluate the hypothesis: Can PEM Flex Solo II PET scanner ascertain response to neoadjuvant chemotherapy in patients with breast cancer?
2. To compare the results from the PEM Flex Solo II PET scanner to the standard of care bilateral breast MRI.

DETAILED DESCRIPTION:
Subjects will receive bilateral (both sides) breast and axillary PEM scans. All recruited subjects chosen for the study will have biopsy proven breast cancer and are eligible for chemotherapy. They will undergo bilateral breast MRI for staging which is considered standard of care. Breast MRI and PEM scans will be performed at at baseline (phase 0 or pre-operative phase), 2nd MRI and PEM after 1 to 2 weeks of NAC (phase 1) and 3rd MRI and PEM after 1 to 2 weeks of phase 1 (phase 2). DCE-MRI and PEM will be performed not more than 14 days apart within each phase. Cranio-Caudal (CC) and Medial Lateral Oblique (MLO) PEM views will be performed of both the ipsilateral and contralateral breast and axillae by a Mammography Technologist trained in mammographic positioning.

ELIGIBILITY:
Inclusion Criteria:

* Women 18-75 years old with newly diagnosed breast cancer who are considered candidates for breast conserving surgery (i.e., lumpectomy)

Exclusion Criteria:

* Children (< 18 years old)
* Pregnant or Lactating women
* Diabetic patients (Type I or II)
* Patients who are scheduled for a sentinel node procedure using radioactive Tc-99m within 24 hours of PEM
* Patients who have NOT undergone a standard of care bilateral breast MRI

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-11; Primary Completion 2011-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kirti Kulkarni, M.D., Principal Investigator — The University of Chicago Medical Center
Locations (1):
- The University of Chicago Medical Center, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Beast Cancer Subjects
Started | 5
Completed | 3
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Beast Cancer Subjects
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (6.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Tumor Size
Description: Comparison of tumor size pre chemotherapy and post chemotherapy represents the PEM data. There is no the response with MRI because the study was aborted and very few patients were involved.
Time Frame: 1-2 weeks post treatment onset
Population: This study has been terminated due to poor accrual.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Beast Cancer Subjects
Number analyzed (Participants) | 3
mm
  PEM tumor size pre chemotherapy | 25.67 (7.5)
  PEM tumor size post chemotherapy | 9.67 (16.7)

ADVERSE EVENTS:
Arm/Group | Beast Cancer Subjects
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes